CLINICAL TRIAL: NCT02556606
Title: Ketamine for Treatment Resistant Late-Life Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLNA-001-14F
Record Dates: First submitted 2015-06-25; First posted 2015-09-22 (Estimated); Results first posted 2021-08-09 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Treatment Resistant Depressive Disorder
Keywords: ketamine; depression; treatment resistant; treatment resistant depression; late life depression; depression in the elderly; geriatric depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: We use a Bayesian, adaptive, randomized design initially allocating subjects to 2 arms in a 1:3 ratio: ARM 1: MID 0.03 mg/kg (active placebo); ARM 2: four conditions KET 0.1 mg/kg, KET 0.25 mg/kg, KET 0.5 mg/kg or MID 0.03 mg/kg. After 1:1:1:1 allocation of the first 20 subjects to ARM 2, Bayesian adaptive randomization may stop for superiority, change randomization ratios and/or prune arms for futility based on the probability of a day 7 treatment response. ARM 1 remains open for allocation to ensure a placebo group sufficiently large for comparison with best dose KET. For analyses, MID of ARM 1 and ARM 2 will be combined so that there are 4 conditions (or arms) for final statistical analyses. We expected to enroll a maximum 72 patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ketamine 0.10 mg/kg (Experimental): randomly assigned to a single 40 min infusion of either KET 0.1mg/Kg
  Interventions: Drug: Ketamine
- Ketamine 0.25 mg/kg (Experimental): randomly assigned to a single 40 min infusion of either KET 0.25mg/Kg
  Interventions: Drug: Ketamine
- Ketamine 0.50 mg/kg (Experimental): randomly assigned to a single 40 min infusion of either KET 0.50mg/Kg
  Interventions: Drug: Ketamine
- Midazolam 0.03 mg/kg (Active Comparator): randomly assigned to a single 40 min infusion of either MID 0.03mg/Kg
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — randomly assigned to a single 40 min infusion of either KET 0.1mg/Kg
  Arms: Ketamine 0.10 mg/kg
Drug: Ketamine — randomly assigned to a single 40 min infusion of either KET 0.25mg/Kg
  Arms: Ketamine 0.25 mg/kg
Drug: Ketamine — randomly assigned to a single 40 min infusion of either KET 0.50mg/Kg
  Arms: Ketamine 0.50 mg/kg
Drug: Midazolam — single 40 min infusion of MID 0.03mg/Kg
  Arms: Midazolam 0.03 mg/kg

SUMMARY:
The purpose of this study is to examine the effectiveness of a single infusion of ketamine (KET), to determine which dose is optimal 7 days after infusion using Bayesian Adaptive Randomization, and to learn about how ketamine works in the body and brain in persons with late-life treatment resistant depression.

DETAILED DESCRIPTION:
Primary Aim: To identify the best performing condition across a single intravenous infusion of ketamine (KET) 0.1 mg/kg, KET 0.25 mg/kg, KET 0.50 mg/kg) and midazolam (MID) 0.03 mg/kg on Montgomery-Asberg Depression Rating Scale (MADRS) treatment response (at least a 50% improvement in depression from baseline) 7 days after the infusion in up to 72 Veterans with Late-Life Treatment Resistant Depression (LL-TRD) , using a triple blind (patient, rater, anesthesiologist) Bayesian adaptive randomization design.

Hypothesis 1: Single KET 0.5 mg/kg infusion is superior to KET 0.1 mg/kg, KET 0.25 mg/kg, and MID 0.03 mg/kg measured by the proportion of participants demonstrating > 50% reduction on MADRS scores 7 days post-treatment.

Secondary Aim: To evaluate the durability of day 7 treatment response across 3 sub-anesthetic doses of a single KET (0.1 mg/kg, 0.25 mg/kg, and 0.50 mg/kg) and MID (0.03 mg/kg) infusion in veterans with LL-TRD during a 4 week follow-up.

Hypothesis 2: a single KET 0.5 mg/kg infusion will be superior to a single infusion of KET 0.1 mg/kg, KET 0.25 mg/kg, and MID 0.03 mg/kg as measured by the proportion of participants demonstrating > 50% reduction on MADRS scores at 28 days post-infusion.

Tertiary Aim: To evaluate the immediate and longer-term safety and tolerability of the most effective KET infusion relative to MID in vets with LL-TRD.

Hypothesis 3: KET infusion at the most effective dose will be safe and well tolerated compared to MID, as assessed by psychoactive and general side effect rating scales during and up to 4 weeks post study infusion.

Exploratory Aims:

1. To measure the effects of the most effective dose of KET relative to MID on neurocognitive performance.
2. To measure the effects the most effective dose of KET relative to MID on peripheral biomarkers of cellular plasticity and inflammation.
3. To measure the effects the most effective dose of KET relative to MID on resting-state quantitative electroencephalography.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 55 years of age,
* Participants must fulfill DSM 5 criteria for a Major Depressive Episode (Unipolar), based on a structured diagnostic interview, the DSM 5 M.I.N.I. 7.0
* Participants must have a history of at least one previous episode of depression prior to the current episode (recurrent MDD) or have chronic MDD (of at least two years' duration),
* Participants have not responded to two or more adequate trials of FDA-approved antidepressants, determined by Antidepressant Treatment Response Questionnaire (ATRQ) criteria.
* Participants must score 14 or greater on the Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR), and score 27 on the Montgomery Asberg Depression Rating Scale (MADRS),
* Each participant must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document.

Exclusion Criteria:

* Patients currently on fluoxetine,
* History of schizophrenia, schizoaffective disorder or any psychotic disorder, or bipolar disorder,
* Documented history of a psychotic disorder in a first-degree relative,
* Current diagnosis of obsessive-compulsive disorder (OCD) or eating disorder [bulimia nervosa or anorexia nervosa],
* Alcohol or substance use [except nicotine] within the preceding 6 months,
* Patients with any clinically significant personality disorder that would, in the investigator's judgment, preclude safe study participation,
* Patients judged to be at serious and imminent suicidal or homicidal risk,
* Serious, unstable medical illnesses including respiratory [obstructive sleep apnea, or history of difficulty with airway management during previous anesthetics], cardiovascular [including ischemic heart disease and uncontrolled hypertension], and neurologic [including history of severe head injury],
* For study entry, patients must be reasonable medical candidates for ketamine or midazolam infusion, as determined by a board-certified physician co-investigator during study Screening,
* Clinically significant abnormal findings of laboratory parameters [including urine toxicology screen for drugs of abuse], physical examination, or ECG,
* Hypertension (systolic BP >160 mm Hg or diastolic BP >90 mm Hg),
* Patients with one or more 11 seizures without a clear and resolved etiology,
* Patients starting hormonal treatment (e.g., estrogen) in the 3 months prior to Screening,
* Past intolerance or hypersensitivity to ketamine, or history of recreational use of phencyclidine (PCP) or ketamine,
* Past intolerance or hypersensitivity to midazolam,
* Age-related cognitive decline or mild dementia suggested by a score of < 25 on the Mini-Mental State Examination (MMSE) at Screening,
* Patients taking medications with known activity at the N-methyl-D-aspartate receptor (NMDA) or AMPA glutamate receptor [e.g., riluzole, amantadine, lamotrigine, memantine, topiramate, dextromethorphan, D-cycloserine], or the muopioid receptor,
* Patients taking any of the following medications: St John's Wort, theophylline, tramadol, metrizamide,
* Patients who demonstrate > 25% decrease in depressive symptoms as reflected by the QIDS-SR score from Screening to Randomization,
* Patients who have received electroconvulsive therapy (ECT) in the past 6 months prior to Screening,
* Patients currently receiving treatment with vagus nerve stimulation (VNS) or repetitive transcranial stimulation (rTMS).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Mathew, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy N, Lijffijt M, Ramakrishnan N, Vo-Le B, Vo-Le B, Iqbal S, Iqbal T, O'Brien B, Smith MA, Swann AC, Mathew SJ. Does mismatch negativity have utility for NMDA receptor drug development in depression? Braz J Psychiatry. 2022 Jan-Feb;44(1):61-73. doi: 10.1590/1516-4446-2020-1685. PMID 33825765

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine 0.10 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.50 mg/kg | Midazolam 0.03 mg/kg
Started | 4 | 5 | 11 | 13
Completed | 4 | 5 | 11 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ketamine 0.10 mg/kg: randomly assigned to a single 40 min infusion of KET 0.1 mg/kg
- Ketamine 0.25 mg/kg: randomly assigned to a single 40 min infusion of KET 0.25 mg/kg
- Ketamine 0.50 mg/kg: randomly assigned to a single 40 min infusion of KET 0.50 mg/kg
- Midazolam 0.03 mg/kg: randomly assigned to a single 40 min infusion of MID 0.03 mg/kg
- Total: Total of all reporting groups
Arm/Group | Ketamine 0.10 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.50 mg/kg | Midazolam 0.03 mg/kg | Total
Number analyzed (Participants) | 4 | 5 | 11 | 13 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.75 (5.54) | 61.8 (6.06) | 60.91 (4.97) | 62.15 (5.54) | 62.24 (5.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 4 | 10
  Male | 4 | 2 | 8 | 9 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 4 | 4 | 11 | 12 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 4 | 7 | 16
  White | 2 | 2 | 7 | 6 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Demonstrating at Least a 50% Reduction on Montgomery-Asberg Depression Rating Scale Scores
Description: To determine the best performing intervention among three sub-anesthetic doses of a single ketamine (0.1 mg/kg, 0.25 mg/kg, and 0.50 mg/kg) and midazolam (0.03 mg/kg) in Veterans with LL-TRD as measured by the percentage of participants demonstrating at least a 50% reduction from pre-treatment baseline on Montgomery-Asberg Depression Rating Scale (MADRS; score range 0 - 60, higher scores meaning more severe depression) scores at 7 days post-infusion.
Time Frame: Day 7 post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine 0.10 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.50 mg/kg | Midazolam 0.03 mg/kg
Number analyzed (Participants) | 4 | 5 | 11 | 13
Participants | 0 | 2 | 8 | 6

2. Secondary Outcome: Percentage of Patients With Continuation From Day 7 to Day 28 Post-infusion of at Least a 50% Improvement in MADRS
Description: Patients with a day 7 treatment response (at least a 50% improvement from baseline in Montgomery-Asberg Depression Rating Scale [MADRS]) are followed until day 28 post-infusion; day 7 non-responders are not followed. Outcome measure is the percentage of patients who continue to be responder at day 28, and is interpreted as a measure of durability of efficacy.
Time Frame: 28 days post-infusion follow-up
Population: Day 7 responders were followed until day 28 post-infusion or until relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine 0.10 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.50 mg/kg | Midazolam 0.03 mg/kg
Number analyzed (Participants) | 0 | 2 | 8 | 6
Participants | 0 | 1 | 7 | 4

3. Other Pre Specified Outcome: Change in Clinician-Administered Dissociative States Scale (CADSS)
Description: Change from pre-infusion baseline to end of infusion at 40 minutes after start of infusion on the Clinician-Administered Dissociative States Scale (CADSS; scale form 0 [no psychosis-like symptoms] to 90 [severe psychosis-like symptoms]) to assess psychosis-like side effect on day of infusion.
Time Frame: Baseline to 40 minutes after start of infusion
Measure: Mean (Standard Deviation); unit: Score on CADSS scale
Arm/Group | Ketamine 0.10 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.50 mg/kg | Midazolam 0.03 mg/kg
Number analyzed (Participants) | 4 | 5 | 11 | 13
Score on CADSS scale
  Pre-infusion baseline | 1.41 (0.71) | 0 (0) | 0.09 (0.30) | 0.23 (0.60)
  End of infusion at 40 minutes | 4.79 (2.39) | 14.98 (6.70) | 21.36 (20.53) | 4.38 (6.73)

4. Other Pre Specified Outcome: Change in Resting-state Quantitative Electroencephalography (EEG) Frontal Gamma Band Power (Log of Microvolt Squared)
Description: Change in EEG frontal gamma power from pre-infusion baseline to 30 minutes after start of infusion to assess engagement of the study drug with the N-methyl-D-aspartate receptor.
Time Frame: Baseline to 30 minutes after start of infusion
Population: Missing data due to poor data quality for KET 0.1 (n=1), KET 0.5 (n=3) or MID (n=3)
Measure: Mean (Standard Deviation); unit: uV^2
Arm/Group | Ketamine 0.10 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.50 mg/kg | Midazolam 0.03 mg/kg
Number analyzed (Participants) | 3 | 5 | 8 | 10
uV^2
  Pre-infusion baseline | 0.0019 (0.0004) | 0.055 (0.0030) | 0.0042 (0.0026) | 0.0061 (0.0078)
  30 minutes after start of infusion | 0.0035 (0.0012) | 0.0057 (0.0044) | 0.0098 (0.0067) | 0.004 (0.0027)

5. Other Pre Specified Outcome: Change in Systolic Blood Pressure (Millimeters of Mercury, mm Hg)
Description: Change in systolic blood pressure from pre-infusion baseline to 30 minutes after start of infusion
Time Frame: Baseline to 30 minutes after start of infusion
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Ketamine 0.10 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.50 mg/kg | Midazolam 0.03 mg/kg
Number analyzed (Participants) | 4 | 5 | 11 | 13
mm Hg
  Pre-infusion baseline | 154.25 (5.91) | 142.2 (15.97) | 132.91 (10.56) | 125.54 (213.01)
  30 minutes after start of infusion | 152.75 (12.97) | 148.2 (18.07) | 160.36 (25.94) | 116.62 (15.56)

6. Other Pre Specified Outcome: Change in Diastolic Blood Pressure (Millimeters of Mercury, mm Hg)
Description: Change in systolic blood pressure from pre-infusion baseline to 30 minutes after start of infusion
Time Frame: Baseline to 30 minutes after start of infusion
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Ketamine 0.10 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.50 mg/kg | Midazolam 0.03 mg/kg
Number analyzed (Participants) | 4 | 5 | 11 | 13
mm Hg
  Pre-infusion baseline | 80.5 (7.05) | 74.6 (13.37) | 82.64 (4.72) | 72.23 (9.36)
  30 minutes after start of infusion | 91.25 (14.24) | 82.6 (18.53) | 95.45 (16.01) | 73.54 (12.29)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Ketamine 0.10 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.50 mg/kg | Midazolam 0.03 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/11 | 1/13
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 11/11 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine 0.10 mg/kg (N=4) | Ketamine 0.25 mg/kg (N=5) | Ketamine 0.50 mg/kg (N=11) | Midazolam 0.03 mg/kg (N=13)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — One participant made a suicide attempt four days after midazolam infusion. The event was determined unrelated to the intervention because this participant scored zero on the Columbia Suicide Severity Rating Scale one day before the attempt
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine 0.10 mg/kg (N=4) | Ketamine 0.25 mg/kg (N=5) | Ketamine 0.50 mg/kg (N=11) | Midazolam 0.03 mg/kg (N=13)
Gastrointestinal complaints (Gastrointestinal disorders) | 4 (4) | 4 (4) | 8 (8) | 11 (11) — Using the Patient Reported Inventory of Side Effects (PRISE) as a score of 1 or 2 (mild to moderate adverse event); scores over 2 indicate serious adverse event and are not reported in this section. Collected to day 7 due to smaller sample to day 28.
Cardiac complaints (Cardiac disorders) | 1 (1) | 3 (3) | 4 (4) | 7 (7) — Collected with the Patient Reported Inventory of Side Effects (PRISE)
Skin complaints (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 7 (7) | 9 (9) — Collected with the Patient Reported Inventory of Side Effects (PRISE)
Nervous system complaints (Nervous system disorders) | 4 (4) | 5 (5) | 7 (7) | 11 (11) — Collected with the Patient Reported Inventory of Side Effects (PRISE)
Eye or ear complaints (Eye disorders) | 3 (3) | 5 (5) | 4 (4) | 11 (11) — Collected with the Patient Reported Inventory of Side Effects (PRISE)
Genital or urinary complaints (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 5 (5) | 6 (6) — Collected with the Patient Reported Inventory of Side Effects (PRISE)
Sleep complaints (General disorders) | 4 (4) | 5 (5) | 11 (11) | 13 (13) — Collected with the Patient Reported Inventory of Side Effects (PRISE)
Sexual functioning complaints (Reproductive system and breast disorders) | 3 (3) | 4 (4) | 9 (9) | 12 (12) — Collected with the Patient Reported Inventory of Side Effects (PRISE)
Other complaints (General disorders) | 4 (4) | 5 (5) | 11 (11) | 13 (13) — Collected with the Patient Reported Inventory of Side Effects (PRISE)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT02556606/Prot_SAP_000.pdf